CLINICAL TRIAL: NCT03775902
Title: Regulation of KATP Channels and Na+/K+ ATPase in Relation to Fatigue Development in Healthy and Insulin Resistant Subjects
Brief Title: Regulation of KATP Channels and Na+/K+ ATPase in Relation to Fatigue Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: NAK-KATP
Record Dates: First submitted 2018-12-04; First posted 2018-12-14 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Insulin Resistance
Keywords: skeletal muscle; muscle fatigue; ion handling
MeSH Terms: conditions — Insulin Resistance | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy subjects (Experimental): Two experimental day where the effect of Nicorandil (20mg) or placebo will asses the function of the ATP sensitive potassium pumps role in the development of fatigue.
  Interventions: Drug: Placebo; Drug: Nicorandil
- Insulin resistant (Experimental): Two experimental day where the effect of Nicorandil (20mg) or placebo will asses the function of the ATP sensitive potassium pumps role in the development of fatigue.
  Interventions: Drug: Placebo; Drug: Nicorandil

INTERVENTIONS:
Drug: Placebo — placebo tablet
Drug: Nicorandil — 20 mg nicorandil (Ikorel, Sanofi Winthrop Industrie; NIC)

SUMMARY:
To investigate the role of ATP sensitive K+ potassium channels and the Na+/K+ pump in the development of fatigue in healthy and in insulin resistant subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non smokers
* HbA1c <38 mmol/mol (<5.7%), HOMA-IR > 1.7 (insulin resistant)
* VO2max <40 ml/kg/min (insulin resistant), 45-55 ml/kg/m2 (healthy)
* BMI >26 kg/m2 (insulin resistant), 19-26 kg/m2 (healthy)

Exclusion Criteria:

* Use of antidiabetic medication or any other medication deemed to interfere with study outcomes
* Allergy towards Nicorandil
* Chronic disease other than type 2 diabetes deemed to interfere with study outcomes
* Excessive alcohol consumption (>14 units/week)
* Abnormal ECG

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Extracellular potassium concentration meassured with microdialysis | Changes in potassium handling from the placebo experimental day compared to the experimental days with Nicorandil ingestion with 14 days between each experimental day. Timeframe pr. subject approx. 6 weeks
  Interstitial potassium

SECONDARY OUTCOMES:
Performance (time to exhaustion) during knee extensor exercise | Changes in performance during the placebo experimental day compared to the experimental days with Nicorandil ingestion with 14 days between each experimental day. Timeframe pr. subject approx. 6 weeks.
  Muscle exercise tolerance

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Copenhagen, Danmark, Denmark